CLINICAL TRIAL: NCT06190015
Title: Impact of Advanced Platelet Rich Fibrin and Enamel Matrix Derivative on Clinical and Molecular Wound Healing Parameters After Surgical Removal of Mandibular Third Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Ruzica Brajovic, principal investigator, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1/36/20
Record Dates: First submitted 2023-12-16; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Surgical Wound, Healed; Post Operative Pain
Keywords: third molar; wound healing; postoperative pain, edema
MeSH Terms: conditions — Surgical Wound; Pain, Postoperative; Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Advanced platelet rich fibrin (APRF) group; (Active Comparator): After surgical removal of one of the impacted mandibular third molar, APRF clots will be placed in the alveolus
  Interventions: Biological: Advanced platelet rich fibrin (APRF) clots
- Control group 1; (No Intervention): Standard surgical removal of the other impacted mandibular third molar will be performed without placing APRF in the wound
- Enamel matrix derivative (EMD) group; (Active Comparator): After surgical removal of one impacted mandibular third molar, EMD with collagen sponges will be placed in the extraction alveolus
  Interventions: Device: Enamel matrix derivative (EMD) group
- Control group 2; (No Intervention): Standard surgical removal of the other impacted mandibular third molar will be performed without placing EMD in the wound

INTERVENTIONS:
Biological: Advanced platelet rich fibrin (APRF) clots — 15 minutes before surgery, phlebotomy will be performed and two vacutainers containing 10ml of blood will be placed in the centrifuge for 8 min and 200g. Acquired APRF clots will be placed in the extraction alveolus
  Arms: Advanced platelet rich fibrin (APRF) group;
Device: Enamel matrix derivative (EMD) group — After third molar removal, Pref Gel (EDTA) will be placed on the root surface for 2 min and then removed. Emdogain (EMD) will be placed on the collagen sponge (Botiss, Collacone) and then applied in the wound so that the side of the sponge which is covered with Emdogain is in contact with the root surface.
  Other Names: Emdogain, Straumann,
  Arms: Enamel matrix derivative (EMD) group;

SUMMARY:
Brief summary

The goal of this study is to compare the effects of advanced platelet rich fibrin and enamel matrix derivative placed in the extraction alveoli of patients who had surgical removal of mandibular wisdom teeth. The questions it aims to answer/evaluate are:

* postoperative pain, swelling, trismus, early wound healing using soft tissue healing index
* level of early local inflammatory response by measuring levels of inflammatory mediators in wound exudate
* degree of wound healing by measuring levels of early wound healing mediators in wound exudate
* incidence of alveolar osteitis and delayed infection
* levels of probing depth, clinical attachment loss, gingival margin level, bleeding on probing, gingival index, plaque index of the second mandibular molar 3 months after surgery

Participants of the study will be asked:

* for their preoperative clinical measurements (swelling, trismus, periodontal parameters) to be taken by the principal investigator
* to provide 20 ml of venous blood if necessary
* to preoperatively provide gingival crevicular fluid in the region of distal surface of the second mandibular molar and postoperatively wound exudate
* to note the number of painkiller pills taken after surgery and pain levels in different time points
* to come to regular checkups in which clinical measuring of postoperative swelling, trismus levels and periodontal parameters will be performed

DETAILED DESCRIPTION:
Surgical removal of impacted mandibular wisdom teeth is often related to the occurrence of postoperative pain, swelling, trismus and sometimes to the development of complications such as alveolar osteitis, delayed infection and formation of periodontal pocket on the distal surface of the second molar. In order to reduce postoperative discomfort and complications, nonsteroidal anti-inflammatory drugs and antibiotics are being routinely prescribed.

Placement of autologous materials and commercially available products in the extraction alveoli, in order to minimize postoperative pain, swelling, trismus and complications, is a therapy option that is discussed in literature.

Platelet rich fibrin (PRF) is an autologous fibrin derived from patient's venous blood rich in platelets, leucocytes, growth factors and cytokines. Advanced PRF (APRF) is a variant of PRF which is produced by smaller centrifugation speed and smaller relative centrifugal force for a longer time period in comparison to the other types of PRF clots. APRF contains leucocytes, vascular endothelial growth factor (VEGF), transforming growth factor β (TGF-β), interleukin -1β (IL1β) and interleukin-6 (IL6).

Local application of APRF in the extraction alveolus after surgical removal of impacted mandibular wisdom teeth has shown positive effects such as lesser postoperative pain, better soft tissue healing and lower incidence of alveolar osteitis and delayed infection.

In vitro studies have shown that PRF contains significant amounts of VEGF, TGF-β, IL1β, IL6. In vitro study also showed that PRF induces polymerization of M1 proinflammatory macrophages to M2 anti-inflammatory macrophages. M2 macrophages produce specialized pro-resolving lipid mediators which are important for resolution phase of inflammatory process and wound healing. Maresin 1 (MaR1), specialized pro-resolving lipid mediator, has shown an important role in inducing faster soft tissue and bone healing and therefore the presence of this mediator may be relevant to indicate the course of postoperative wound healing. Taking into consideration the data from clinical and in vitro studies, it would be beneficial to determine on a clinical model such as surgical removal of impacted mandibular wisdom teeth levels of VEGF, TGF-β, IL1β, IL6 and MaR1 after placing APRF into the extraction alveolus in comparison to the standard surgical removal of impacted mandibular wisdom teeth and compare those levels with clinical parameters of postoperative course.

Enamel matrix derivative (EMD) contains enamel matrix proteins amelogenins extracted from six-month-old piglets. Cells of the Hertwig's epithelial root sheath release predominantly amelogenins on the root surface prior to cementum formation, and these proteins are the initiating factor for cementogenesis during odontogenesis. In vitro studies have shown that periodontal ligament cells exposed to EMD produce TGF-β and IL6. Similar study has shown that the expresion of IL1β was significantly lower after exposure of periodontal ligament cells to the EMD. Clinical and in vitro study have shown that EMD stimulates angiogenesis by inducing human microvascular endothelial cells to produce VEGF. Positive influence of EMD on periodontal defects is shown by many clinical studies.

Regarding clinical and in vitro studies, significant levels of VEGF, TGF-β, IL1β, IL6 after placing EMD could in a clinical model of surgical removal of impacted wisdom teeth indicate better wound healing, periodontal parameters of second molar and lesser postoperative discomfort and complications. In the literature there are no information on potential influence of EMD on production of Mar1.

The primary goal of the research will be to evaluate and compare local inflammatory response and soft tissue healing between the groups where APRF or EMD were placed and standard surgical removal of impacted mandibular wisdom teeth by determining and comparing levels of IL6, IL1β, Mar1, VEGF and TGF-β. Also the primary goal is to evaluate and compare levels of postoperative pain, swelling, trismus and soft tissue healing. Secondary goals are to evaluate incidence of alveolar osteitis, delayed infection and development of periodontal pocket on the distal surface of the lower second molar and analyze between the groups and find out if the correlation between clinical and molecular parameters exists.

A prospective, randomized, controlled, double split mouth study will be conducted at the Department of Oral surgery and Laboratory for basic science, School of Dental medicine, University of Belgrade, Serbia. The research will be performed following the CONSORT guidelines, per the Helsinki Declaration. After meeting the inclusion criteria, participants will receive verbal and written information on the study objectives, protocol as well as the possible risks and benefits of the study. Only the eligible subjects who agree with the information provided and sign an informed consent form will be enrolled in the study. A total of 60 patients (120 operations) with bilaterally impacted mandibular wisdom teeth will be included. Computer-generated blocked randomization with a 1:1 allocation ratio (block size 4) will be performed by a researcher not included in the study (Microsoft Excel, version 2016). To conceal the allocation, the papers containing a code of the allocated group (1-APRF group; 2-EMD group) will be placed in opaque envelopes and sealed. One hour before the intervention, the same independent researcher will unseal the following envelope. After discovering the experimental group (APRF or EMD), the independent researcher will allocate the side of the jaw to the control group or experimental group by flipping a coin.

In the APRF group 15 minutes before the surgery, the independent researcher will inform the patient that phlebotomy will be performed and instruct the phlebotomist to perform the phlebotomy. The principal investigator will be unaware of the allocation until finishing the data analysis. The surgeon will be aware of the allocation due to the nature of the intervention.

Enrollment criteria for the study are systemically healthy patients who have bilaterally impacted mandibular wisdom teeth which are in contact with the distal surface of the second mandibular molar.

Age (years), gender and smoking status (no smoking, ≤10/day, or >10/day) will be obtained from patients who have met the enrollment criteria. At the same appointment (first study appointment), both surgical interventions will be scheduled with at least three weeks apart. Third molar position will be estimated on panoramic radiographs, according to the Pell and Gregory and Winter classifications. Initial exam, perioperative, intraoperative and follow up measurements will be performed by one blinded clinician.

Gingival crevicular fluid sampling on the distal surface of the second mandibular molar , baseline measurements of maximal inter-incisor and distances tragus- oral commissure, outer canthus-angle of the mandible at the side of the extraction and periodontal measuring of the second mandibular molar will be performed at the second study appointment, just before the surgery. Periodontal charting will be performed in three points buccally and in three following points, medial distal, lingual distal, medial lingual point.

After regional inferior alveolar, lingual, and buccal nerve blocks with a local anesthetic solution, consisting of 4% articaine hydrochloride with 1:100000 epinephrine (Septanest ®, Septodont, Saint-Maur-des-Fosses, France), the surgical removal of impacted mandibular third molar will be performed according to the technique previously described in the literature: after full-thickness flap elevation, bone removal will be performed by rotatory instruments under sterile saline irrigation. Elevators and pliers will be used for tooth extraction and tooth separation will be performed, if necessary. After tooth extraction and bone edges smoothening, in the APRF group two APRF clots will be placed in the alveolus and in the EMD group, distal root surface of the second molar will be treated with 24% EDTA (( PrefGel®, Straumann) for two minutes, then irrigated and EMD ( Emdogain®, Straumann) will be placed in combination with collagen sponge ( Collacone®, Botiss). The wound will be sutured with 4-0 polypropylene suture material with special note to place first two consequent sutures in the retromolar region with 5 mm distance in order to allow sampling of wound exudate by placing paper points in the wound at the follow ups.

In control groups after tooth extraction and bone edges smoothening, primary suture will be immediately placed with the same note mentioned before.

All the surgical procedures will be performed by one experienced oral surgeon. Intraoperatively, the duration of the intervention (min), the amount of local anesthetic solution used (ml), tooth separation if performed, and any intraoperative complications will be registered.

Patients will be given paracetamol 500 mg tablets ((Paracetamol®, Galenika, Belgrade, Serbia) to take home and a pre-designed take-home query which contains fields for analgesic registration (every time of intake, number of taken pills and dose). Additionally, patients will be instructed to record pain intensity on visual analog scale (VAS) and verbal rating pain scale (VRS).

At the third study appointment (24h after surgery) measurement of maximal inter-incisor and distances tragus- oral commissure, outer canthus-angle of the mandible at the side of the extraction will be taken. Patients will also be asked to evaluate their pain intensity at the appointment on VAS and VRS.

At the fourth study visit (48h after surgery) maximal inter-incisor measurement and distances tragus- oral commissure, outer canthus-angle of the mandible at the side of the extraction will be taken. In this visit sampling of the wound exudate will also be performed and patients will be asked once again to evaluate their pain level on VAS and VRS.

At the fifth study visit (7 days after surgery), maximal inter-incisor measurement and distances tragus-oral commissure, outer canthus-angle of the mandible will be taken. Also wound exudate sampling will be performed before suture removal. At this visit patients will bring back their previously given query which they have been fulfilling during the week.

The sixth study visit will occur three months after surgery and periodontal charting will be performed.

Samples will be taken by paper points (size #30, 28mm long ISO standardized points with a taper of 2%) placed in the wound for 30s. Measures would be taken to prevent saliva contamination of paper points during sampling. Paper points will be then placed in sterile plastic tubes that are pre-filled with fluid that prevents RNA.

Laboratory procedures will be performed with aim to assess the level of relative gene as well as protein expression of inflammatory (IL6, IL1β, MAR1) and early wound healing (VEGF, TGF-β) mediators in tested groups in different time points of interest. After RNA isolation and obtaining complementary DNA (according to the manufacturer's instructions), relative gene expression of IL6, IL1β,VEGF and TGF-β will be evaluated by means of real-time polymerase chain reaction assay. Protein expression of MAR1 will be performed by enzyme linked immunosorbent assay (ELISA).

Statistical analysis will be performed in statistical package SPSS, version 22.0 (SPSS, Inc. Chicago). Data will be presented through mean, standard deviation, median, maximum and minimum values, percent. Depending of the data distribution, appropriate parametric or non-parametric tests will be performed. Regression models will be performed to determine the predictors of detected inter-group differences. The level of significance will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals (ASA I by American Society of Anesthesiologists classification);
* Age 18-30 years;
* Patients who have bilaterally impacted mandibular wisdom teeth which are in contact with the distal surface of the second mandibular molar.

Exclusion Criteria:

* Systemic disorders;
* Patients who have difficulties when phlebotomy is performed
* History of pericoronitis in the area of impacted mandibular wisdom tooth
* History of NSAIDs, corticosteroids and antibiotics intake within 10 days before surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-01-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of postoperative pain on visual analog scale | 24 hours after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | 24-48 hours after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | 48-72 hours after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | 72 hours- 7 days after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on verbal rating scale | 24 hours after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | 24-48 hours after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | 48-72 hours after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | 72 hours- 7 days after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain by marking the number of pain tablets and time of their consumption | 24 hours after surgery
  After measuring their pain level on VAS and VRS, patients will be writing the number of Paracetamol tablets (500mg) that were taken and exact time of their consumption.
Evaluation of postoperative pain by marking the number of pain tablets and time of their consumption | 24-48 hours after surgery
  After measuring their pain level on VAS and VRS, patients will be writing the number of Paracetamol tablets (500mg) that were taken and exact time of their consumption.
Evaluation of postoperative pain by marking the number of pain tablets and time of their consumption | 48-72 hours after surgery
  After measuring their pain level on VAS and VRS, patients will be writing the number of Paracetamol tablets (500mg) that were taken and exact time of their consumption.
Evaluation of postoperative pain by marking the number of pain tablets and time of their consumption | 72 hours- 7 days after surgery
  After measuring their pain level on VAS and VRS, patients will be writing the number of Paracetamol tablets (500mg) that were taken and exact time of their consumption.
Evaluation of preoperative tragus- oral commissure and outer eye canthus-angle of the mandible distances at the side of the extraction | 1 hour preoperatively
  Postoperative swelling will be evaluated by measuring distances tragus- oral commissure and outer eye canthus-angle of the mandible at the side of the extraction by using soft tape, expressed in millimeters.
Evaluation of postoperative swelling | 24 hours after surgery
  Postoperative swelling will be evaluated by measuring distances tragus- oral commissure and outer eye canthus-angle of the mandible at the side of the extraction by using soft tape, expressed in millimeters.
Evaluation of postoperative swelling | 48 hours after surgery
  Postoperative swelling will be evaluated by measuring distances tragus- oral commissure and outer eye canthus-angle of the mandible at the side of the extraction by using soft tape, expressed in millimeters.
Evaluation of postoperative swelling | 72 hours after surgery
  Postoperative swelling will be evaluated by measuring distances tragus- oral commissure and outer eye canthus-angle of the mandible at the side of the extraction by using soft tape, expressed in millimeters.
Evaluation of postoperative swelling | 7 days after surgery
  Postoperative swelling will be evaluated by measuring distances tragus- oral commissure and outer eye canthus-angle of the mandible at the side of the extraction by using soft tape, expressed in millimeters.
Evaluation of preoperative maximal inter-incisor distance | 1 hour preoperatively
  Maximal inter-incisor distance at baseline will be measured by means of a soft tape, and expressed in millimeters (mm).
Evaluation of postoperative trismus | 24 hours postoperatively
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Evaluation of postoperative trismus | 48 hours postoperatively
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Evaluation of postoperative trismus | 7 days postoperatively
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Relative gene expression of inflammatory and wound healing mediators in gingival crevicular fluid of the distal sulcus of the second mandibular molar preoperatively | 1 hour preoperatively
  To measure the relative gene expression of VEGF, TGF-β1, IL-6, IL-1β in samples of gingival crevicular fluid before surgical removal of impacted mandibular wisdom teeth.
Protein expression of specialized pro-resolving inflammation mediator maresin 1 (Mar1) in gingival crevicular fluid of the distal sulcus of the second mandibular molar preoperatively | 1 hour preoperatively
  To measure the protein expression of Mar1 in samples of gingival crevicular fluid before surgical removal of impacted mandibular wisdom teeth
Relative gene expression of inflammatory and wound healing mediators in wound exudate after surgical removal of impacted mandibular wisdom teeth | 48 hours postoperatively
  To measure the relative gene expression of VEGF, TGF-β1, IL-6, IL-1β in samples of wound exudate after surgical removal of impacted mandibular wisdom teeth.
Relative gene expression of inflammatory and wound healing mediators in wound exudate after surgical removal of impacted mandibular wisdom teeth | 7 days postoperatively
  To measure the relative gene expression of VEGF, TGF-β1, IL-6, IL-1β in samples of wound exudate after surgical removal of impacted mandibular wisdom teeth.
Protein expression of specialized pro-resolving inflammation mediator maresin 1 (Mar1) in wound exudate after surgical removal of impacted mandibular wisdom teeth | 48 hours postoperatively
  To measure the protein expression of Mar1 in samples of wound exudate after surgical removal of impacted mandibular wisdom teeth
Protein expression of specialized pro-resolving inflammation mediator maresin 1 (Mar1) in wound exudate after surgical removal of impacted mandibular wisdom teeth | 7 days postoperatively
  To measure the protein expression of Mar1 in samples of wound exudate after surgical removal of impacted mandibular wisdom teeth.
Evaluation of soft tissue healing using Landry healing index | 7 days after surgery
  Independent researcher will evaluate soft tissue healing by marking the number in front of the given description: 1. Very poor- tissue color: more than 50% of gingivae red Response to palpation: bleeding Granulation tissue: present Incision margin: not epithelialised, with loss of epithelium beyond margins Suppuration: present; 2. Poor- Tissue color: more than 50% of gingivae red Response to palpation: bleeding Granulation tissue: present Incision margin: not epitheliased with connective tissue exposed. 3. Good- Tissue color: less than 50% of gingivae red Response to palpation: no bleeding Granulation tissue: none Incision margin: no connective tissue exposed 4. Very good- Tissue color: less than 25% of gingivae red Response to palpation: no bleeding Granulation tissue: none Incision margin: no connective tissue exposed 5. Excellent-Tissue color: all gingivae pink Response to palpation:no bleeding Granulation tissue:none; Incision margin:no connective tissue exposed

SECONDARY OUTCOMES:
Evaluation of preoperative probing depth of mandibular second molar in six points | 1 hour preoperatively
  Probing depth is the distance from the base of the sulcus/pocket to the gingival margin and it will be measured in three following buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface using periodontal probe calibrated in millimeters. The measurements will be expressed in millimeters.
Evaluation of postoperative probing depth of mandibular second molar in six points | 3 months after surgery
  Probing depth is the distance from the base of the sulcus/pocket to the gingival margin and it will be measured in three following buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface using periodontal probe calibrated in millimeters. The measurements will be expressed in millimeters.
Evaluation of preoperative gingival margin level of mandibular second molar in six points | 1 hour preoperatively
  Gingival margin level is the distance from gingival margin to the cementoenamel junction and it will be measured in three following buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface using periodontal probe calibrated in millimeters. The measurements will be expressed in millimeters.
Evaluation of postoperative gingival margin level of mandibular second molar in six points | 3 month after surgery
  Gingival margin level is the distance from gingival margin to the cementoenamel junction and it will be measured in three following buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface using periodontal probe calibrated in millimeters. The measurements will be expressed in millimeters.
Evaluation of preoperative clinical attachment level of mandibular second molar in six points | 1 hour preoperatively
  Clinical attachment level of mandibular second molar will be evaluated through a formula by subtracting gingival margin level measurement from probing depth measurement in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface. The measurements will be expressed in millimeters.
Evaluation of postoperative clinical attachment level of mandibular second molar in six points | 3 months after surgery
  Clinical attachment level of mandibular second molar will be evaluated through a formula by subtracting gingival margin level measurement from probing depth measurement in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface of second molar, lingual distal point and mid lingual point on the lingual surface. The measurements will be expressed in millimeters.
Evaluation of preoperative bleeding on probing of mandibular second molar in six points | 1 hour preoperatively
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface, lingual distal point and mid lingual point on the lingual surface. Occurrence of bleeding on gentle probing will be marked as 1, no bleeding will be marked as 0.
Evaluation of postoperative bleeding on probing of mandibular second molar in six points | 3 months after surgery
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface, lingual distal point and mid lingual point on the lingual surface. Occurrence of bleeding on gentle probing will be marked as 1, no bleeding will be marked as 0.
Evaluation of preoperative plaque index score of mandibular second molar | 1 hour preoperatively
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface. Each point will be given one of the following scores: 0- no plaque; 1-thin plaque layer at the gingival margin, only detectable by probing; 2-moderate plaque layer at the gingival margin, plaque visible to the naked eye; 3-abundant plaque along the gingival margin, interdental spaces filled with plaque.
  The score will be expressed in the mean value of acquired measurements.
Evaluation of postoperative plaque index score of mandibular second molar | 3 months postoperatively
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface. Each point will be given one of the following scores: 0- no plaque; 1-thin plaque layer at the gingival margin, only detectable by probing; 2-moderate plaque layer at the gingival margin, plaque visible to the naked eye; 3-abundant plaque along the gingival margin, interdental spaces filled with plaque.
  The score will be expressed in the mean value of acquired measurements.
Evaluation of preoperative gingival index score of mandibular second molar | 1 hour preoperatively
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface. Each point will be given one of the following scores: 0-normal gingiva; 1- mild inflammation: slight change in color, slight edema, no bleeding on probing; 2 -moderate inflammation: redness, edema, and glazing or bleeding on probing; 3- severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration.
  The score will be expressed in the mean value of acquired measurements.
Evaluation of postoperative gingival index score of mandibular second molar | 3 months after surgery
  Gentle periodontal probing will be performed in three buccal points, mesial, mid buccal, distal and in medial distal point on the distal surface. Each point will be given one of the following scores: 0-normal gingiva; 1- mild inflammation: slight change in color, slight edema, no bleeding on probing; 2 -moderate inflammation: redness, edema, and glazing, or bleeding on probing; 3- severe inflammation: marked redness and edema, tendency toward spontaneous bleeding, ulceration.
  The score will be expressed in the mean value of acquired measurements.
Incidence of postoperative alveolar osteitis | Within 7 days after surgery
  Occurrence of postoperative complication such as alveolar osteitis will be monitored within first 7 days after surgery and recorded.
Incidence of postoperative infection | Within 3 months after surgery
  Occurrence of postoperative complication such as postoperative infection will be monitored within first three months after surgery and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Snjezana Colic, professor of oral surgery, Study Chair — School of dental medicine, University of Belgrade, Serbia
Locations (1):
- School of dental medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available only to researcher who will enroll the participants and collect the data

REFERENCES:
- [Background] Nasirzade J, Kargarpour Z, Hasannia S, Strauss FJ, Gruber R. Platelet-rich fibrin elicits an anti-inflammatory response in macrophages in vitro. J Periodontol. 2020 Feb;91(2):244-252. doi: 10.1002/JPER.19-0216. Epub 2019 Sep 14. PMID 31376159
- [Result] Gupta N, Agarwal S. Advanced-PRF: Clinical evaluation in impacted mandibular third molar sockets. J Stomatol Oral Maxillofac Surg. 2021 Feb;122(1):43-49. doi: 10.1016/j.jormas.2020.04.008. Epub 2020 Apr 29. PMID 32360489
- See also: This study was conducted on patients who had bilateral impacted third molars. One quadrant received A-PRF while the opposing quadrant in same patient was taken as control. — https://pubmed.ncbi.nlm.nih.gov/32360489/